CLINICAL TRIAL: NCT03865238
Title: A Phase 3, Prospective, Randomized, Double-blind, Placebo-controlled, Multi-region Study to Evaluate the Efficacy, Safety, and Immunogenicity of Inactivated EV71 Vaccine Produced in Vero Cells With Adjuvant in Infants and Children
Brief Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of an EV71 Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-EV-31
Record Dates: First submitted 2019-02-20; First posted 2019-03-06 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2021-06

CONDITIONS: Enterovirus 71 Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EV71vac (Experimental)
  Interventions: Biological: EV71vac
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: EV71vac — Subjects are to receive a 0.5 mL IM injection of EV71vac. Study drug is administered on Day 1 and Day 57 of the study. Subjects 2 months to < 2 years of age will receive a booster vaccination on Day 366.
  Arms: EV71vac
Biological: Placebo — Subjects are to receive a 0.5 mL IM injection of placebo. Study drug is administered on Day 1 and Day 57 of the study. Subjects 2 months to < 2 years of age will receive a booster vaccination on Day 366.
  Arms: Placebo

SUMMARY:
Subjects will receive the first IM injection of study vaccine on Day 1 and will receive a second dose 56 days later. A booster vaccine will be given 365 days after the first dose in subjects 2 months to < 2 years of age. The last study visit is on Day 422 when subjects will be contacted via telephone / home visit system to assess for adverse events and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children and infants aged from 2 months to less than 6 years as established by medical history and clinical examination.
2. The subjects' parents/guardians are able to understand and sign the ICF.

Exclusion Criteria:

1. Age < 2 months or ≥ 6 years.
2. For subjects < 1 year, gestational age < 34 weeks or birth weight < 2200 grams.
3. Has poor venous access (for subjects in sub-study only).
4. Currently has a fever defined as ear/rectal temperature ≥ 38°C or axillary temperature ≥ 37.5 °C within 2 days before the time of planned vaccination.
5. Has had previous known exposure to EV71 or has received EV71 vaccine.
6. Has a history of herpangina or HFMD associated with enterovirus infection in the past 30 days before the date of the planned study drug vaccination.
7. Has been diagnosed with a significant neurological, pulmonary, cardiovascular, hematological, hepatic, or renal disorder.
8. Has a history of hypersensitivity to vaccines, or a history of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
9. Has used any investigational/non-registered product (including drug, vaccine, or invasive medical device) within 28 days before vaccination or plan to use during the study period.
10. Has confirmed or suspected autoimmune disorder, or immunodeficiency.
11. Administration of any licensed live attenuated vaccine within 14 days before or after each study vaccination (with the exceptions of live attenuated Rotavirus vaccine via oral route).
12. Has used immunoglobulins or any blood products within 11 months before vaccination or plan to use during the whole study period.
13. Has had immunosuppressants, cytotoxic drugs, corticosteroids (including prednisolone ≥ 0.5 mg/kg/day or equivalent), or immunomodulators taken for > 14 days within 6 months before first vaccination or plan to use before the last scheduled study visit. (Inhaled and topical steroids are allowed).
14. Has any medical or psychiatric condition, that is a contraindication to protocol participation based on the judgment of the Investigator.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3061 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Laboratory Confirmed EV71-Associated Disease | Approximately 14 months
  The primary outcome is the number of Laboratory confirmed EV71-associated disease by viral isolation or CODEHOP assay.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, MD, Principal Investigator — National Taiwan University Hospital
Locations (6):
- Taiwan (5):
  - Mackay Memorial Hospital, HsincChu, Hsinchu
  - Taichung Veteran General Hospital, Taichung
  - Mackay Memorial Hospital, Taipei, Taipei
  - National Taiwan Univeristy Hospital, Taipei
  - Chang Gung Memorial Hospital, LinKou, Taoyuan District
- Pasteur Institute of HCMC, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Nguyen TT, Chiu CH, Lin CY, Chiu NC, Chen PY, Le TTV, Le DN, Duong AH, Nguyen VL, Huynh TN, Truong HK, Phan TL, Nguyen TTT, Shih SR, Huang CG, Weng YJ, Hsieh EF, Chang S, Chen C, Tai IC, Huang LM. Efficacy, safety, and immunogenicity of an inactivated, adjuvanted enterovirus 71 vaccine in infants and children: a multiregion, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet. 2022 Apr 30;399(10336):1708-1717. doi: 10.1016/S0140-6736(22)00313-0. Epub 2022 Apr 12. PMID 35427481